CLINICAL TRIAL: NCT02762422
Title: Serial Phlebotomy in Voluntary Blood Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Stuart Katz, Principal Investigator, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08-411; 1R01HL086932 (NIH); UL1TR000038 (NIH)
Record Dates: First submitted 2016-05-02; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Atherosclerosis
Keywords: endothelial function; iron stores; red blood cell; blood donation
MeSH Terms: conditions — Atherosclerosis | interventions — Phlebotomy; Blood Donation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phlebotomy plus normal saline (Experimental): Four serial phlebotomy procedures followed by infusion of normal saline
  Interventions: Other: Phlebotomy
- Phlebotomy plus intravenous iron (Experimental): Four serial phlebotomy procedures followed by infusion of intravenous iron sucrose
  Interventions: Other: Phlebotomy
- Sham Phlebotomy (Placebo Comparator): Four serial sham phlebotomy procedures followed by infusion of normal saline
  Interventions: Other: Phlebotomy

INTERVENTIONS:
Other: Phlebotomy — Removal of 500 cc of blood via forearm vein
  Other Names: Blood donation

SUMMARY:
Blood donation has been proposed to be associated with reduced risk of cardiovascular disease, but the effects of phlebotomy on vascular function in human subjects have not been well characterized. A prospective randomized double-blind study was undertaken to determine the effects of iron loss and red blood cell loss induced by serial phlebotomy on vascular endothelial function in the brachial artery.

DETAILED DESCRIPTION:
84 Fe-replete, non-anemic subjects were randomly assigned to one of three experimental serial phlebotomy procedures designed to induce Fe loss or RBC loss. Brachial artery reactivity (BAR, %) in response to transient oxidative stress induced by oral methionine was measured with high-resolution duplex ultrasound imaging before and after study phlebotomy procedures.

ELIGIBILITY:
Inclusion Criteria:

* hemoglobin levels >13.5 g/dl for men, or >12.5 g/dl for women
* serum ferritin 50-400 ng/ml

Exclusion Criteria:

* known intolerance of phlebotomy procedures
* major trauma or surgical procedures in the last 2 years
* menstrual or other uterine bleeding in the last 2 years
* chronic oral anticoagulation or dual antiplatelet therapy
* chronic non-steroidal anti-inflammatory drug use
* known history of hemochromatosis or other disorder of hematopoiesis or Fe metabolism
* chronic oral Fe supplementation other than Fe-containing multivitamins
* history of active cancer in the past 2 years
* known history of chronic inflammatory disease
* uncontrolled hypertension
* electrocardiographic evidence of prior myocardial infarction
* diabetes mellitus
* fasting glucose >100 mg/dL
* body mass index >40 kg/m2
* any tobacco use in the past 6 months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Brachial artery reactivity response to oral methionine administration | Before and 1 week after completion of assigned phlebotomy procedures
  Measure by vascular ultrasound imaging

SECONDARY OUTCOMES:
Iron deficiency anemia | before each phlebotomy procedure, and at 1, 8, and 16 weeks after completion of assigned phlebotomy procedures
  hemoglobin level measured by hemocue or complete blood count

OTHER OUTCOMES:
Serum ferritin | Before and 1 week after completion of assigned phlebotomy procedures
Serum nitrotyrosine | Before and 1 week after completion of assigned phlebotomy procedures
Whole blood viscosity | Before and 1 week after completion of assigned phlebotomy procedures

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
PI will make de-identified dataset available upon request in accord with institutional data use agreement policy